CLINICAL TRIAL: NCT02939274
Title: An Open Label, Phase II Trial of Continuous Low-Irradiance Photodynamic Therapy (CLIPT) Using Verteporfin (Visudyne®) for the Treatment of Cutaneous Metastases of Breast Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Rogers Sciences Inc. (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RSI-CLIPT-002
Record Dates: First submitted 2016-10-18; First posted 2016-10-20 (Estimated); Last update posted 2018-07-20 (Actual); Status verified 2018-07

CONDITIONS: Metastatic Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Verteporfin

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Open Label (Other): Continuous Low-Irradiance Photodynamic Therapy (CLIPT) Using Verteporfin
  Interventions: Drug: Verteporfin; Device: Continuous Low-Irradiance Photodynamic Therapy (CLIPT)

INTERVENTIONS:
Drug: Verteporfin
Device: Continuous Low-Irradiance Photodynamic Therapy (CLIPT)
  Other Names: CLIPT Illumination System

SUMMARY:
The purpose of this Phase II study is to evaluate the efficacy and safety of Continuous Low- Irradiance Photodynamic Therapy (CLIPT) when used with Verteporfin in the treatment of cutaneous metastases of breast cancer for which no curative or significantly palliative therapy exists, including chest wall therapy.

ELIGIBILITY:
Inclusion Criteria:

* Histologically or cytologically confirmed Stage IIIb or IV breast cancer with cutaneous metastases.

Exclusion Criteria:

* Participants receiving any medications or substances that are known to cause photosensitivity (e.g. tetracyclines, sulfonamides, phenothiazines, sulfonylurea hypoglycemic agents, thiazide diuretics, griseofulvin, fluoroquinolones, St. Johns' wort, amiodarone) are ineligible.
* Participants who have received prior systemic therapy (chemotherapy or targeted therapy) within 7 days of Study Day 1 or those who have not recovered from clinically significant adverse events due to agents administered more than 7 days earlier. (continuation of the same regimen of HER-2 antibody targeted therapy agents, hormonal therapy and treatment with bisphosphonates or denosumab are permitted)
* Participants who are receiving any other investigational agents during the proposed treatment cycle.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Estimated)
Dates: Start 2016-10; Primary Completion 2018-12 (Estimated); Study Completion 2019-12 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate | Day 23
  To evaluate the objective response rate (ORR=CR+PR) at Day 23 (3 weeks) after the initial treatment. The objective response rate is defined as the rate of complete response (CR) plus the rate of partial response (PR).

CONTACTS AND LOCATIONS:
Overall Officials: Steven J Isakoff, MD PhD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Dana Farber Cancer Institute, Boston, Massachusetts